CLINICAL TRIAL: NCT03205241
Title: Effect of 4 Weeks Fish Oil Supplementation on Cycling Performance or Oxidative and Inflammatory Parameters in Healthy Male Cyclists
Brief Title: Effect of 4 Weeks Fish Oil Supplementation on Cycling Performance in Healthy Male Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Worcester (Other)
Responsible Party: Principal Investigator, Lynsey Wilson, Technical Tutor in Exercise Physiology, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R14-P72
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Exercise-induced Inflammation
Keywords: Exercise; Fish Oil; Cycling; Inflammation; Oxidative stress
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double blind, crossover design study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3 PUFA (Experimental): Omega-3 polyunsaturated fatty acid - 5.7g/ day for 4 weeks
  Interventions: Dietary Supplement: n-3 PUFA
- Placebo (Placebo Comparator): Olive Oil - 6g/ day for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 PUFA — n-3 PUFA capsules containing EPA and DHA
  Other Names: Fish Oil supplementation; Omega-3
  Arms: n-3 PUFA
Dietary Supplement: Placebo — Olive oil capsules
  Other Names: Olive Oil
  Arms: Placebo

SUMMARY:
Research Plan

Eleven trained cyclists have completed 4 cycling performance trials, before and after 4 weeks of fish oil supplementation and before and after 4 weeks of placebo with a 4 week washout between supplementation periods. During the performance trials blood, expired air and heart rate were collected. The blood samples have been used to investigate the production of inflammation resulting from the cycling performance test. Inflammation has been assessed using enzyme-linked immunosorbent assay for IL-6, which is an inflammatory cytokine. Work done from the cycling performance will be analysed to investigate whether there is a relationship with power and inflammation and whether this is modulated by fish oil supplementation.

Specific Aims

1. Does 4 weeks of Fish Oil supplementation attenuate the inflammatory response following high intensity cycling.
2. Is a modulation of the inflammatory response connected to cycling performance.

Hypotheses

1. Four weeks of n3-PUFA supplementation will reduce the inflammatory response
2. A reduction in inflammation will improve cycling performance

Anticipated Outcomes

A high level of cycling performance, indicated by a high average power, will be associated with high levels of systemic inflammation. n3-PUFA supplementation will decrease the level of inflammation and consequently cycling performance will be improved.

ELIGIBILITY:
Inclusion Criteria:

* recreationally trained male cyclists

Exclusion Criteria:

* History of coagulation/bleeding disorder
* History of metabolic disease
* Serious allergy
* History of heart disease
* Regular use of anti-inflammatory drugs
* Vitamin or fish oil supplementation over the past 6 months
* Known to have blood-borne virus
* Females

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Work Done | 15 minutes during time trial
  Work done measured in Joules from the Lode cycle ergometer during 15 minute cycling time trial

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey S Wilson, MSc, Principal Investigator — Loughborough University

IPD SHARING:
Plan to Share IPD: No